CLINICAL TRIAL: NCT04253717
Title: Effects of a Motor Control Exercise Program on Lumbopelvic Pain Occurrence and Intensity in Pregnant Women With a History of Lumbopelvic Pain: a Study Protocol for a Randomized Controlled Feasibility Trial.
Brief Title: Motor Control Exercise Program for Pregnant Women With a History of Lumbopelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Trois-Rivières (Other)
Responsible Party: Principal Investigator, Martin Descarreaux, Principal investigator, Université du Québec à Trois-Rivières
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UQTR-2019-LBPP-Intervention
Record Dates: First submitted 2020-01-28; First posted 2020-02-05 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Lumbopelvic Pain
Keywords: Physical activity; Non-invasive treatment
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor control exercise program (Experimental): Participants will be physically trained during pregnancy and will receive the standard care including basic information on what to do when suffering from lumbopelvic pain.
  Interventions: Other: Motor control exercise program
- Control (No Intervention): Participants will receive the standard care including basic information on what to do when suffering from lumbopelvic pain.

INTERVENTIONS:
Other: Motor control exercise program — Structure physical training aimed at strengthening muscles of the lumbo-pelvic-hip core complex in order to improve stabilization and alignment of the spine and pelvis.
  Arms: Motor control exercise program

SUMMARY:
This study protocol was designed to establish the feasibility of conducting a motor control exercise program with pregnant women presenting a history of lumbopelvic pain (LBPP) in order to reduce LBPP occurrence or limit its intensity. This randomized controlled trial also aims to preliminary assess the effectiveness of the program. To do so, 40 pregnant women with a history of LBPP will be recruited and randomly allocated to one of 2 groups: control (20 participants) or intervention (20 participants). The control group will receive standard care, including basic information on what to do when suffering from LBPP. The intervention group will participate in a weekly 40-minute group session and two more 40-minute weekly home exercise sessions. The motor control exercise program will be designed to target strengthening of the lumbo-pelvic-hip core muscles in order to improve stabilization and protection of the spine and pelvis. Participants of this group will also receive standard care. Adequate prevention and treatment of LBPP, experienced by women during pregnancy, should help reduce LBPP occurrence or limit its intensity during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Being pregnant of one fetus
* Being ≤ 20 weeks pregnant
* Presenting a history of lumbopelvic pain

Exclusion Criteria:

* Inflammatory rheumatic disease
* Infectious disease
* Neuromuscular disease
* Vascular disease
* Connective tissue disease
* Severe disabling pain
* Neurologic signs and symptoms

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Baseline (Pre-intervention)
  Defined as the ability to recruit 40 eligible women, willing to participate to the study
Retention rate | Baseline (Post-intervention)
  Defined as the completion of follow-up questionnaire by ≥ 80% of women
Adherence rate | Baseline (Post-intervention)
  Defined as attendance to ≥75% of group sessions and ≥ 75% completion of home sessions
Safety of the intervention | 16 weeks follow-up
  Determined based on the number of adverse events and defined as nature of adverse events
Safety of the intervention | Week 16 (Post-intervention)
  Determined based on the number of adverse events and defined as nature of adverse events
Acceptability of the intervention | 16 weeks follow-up
  Determined based on how the intervention is perceived by pregnant women (assessed using a 5-point Likert scale : higher score mean a better outcome)
Acceptability of the intervention | Week 16 (Post-intervention)
  Determined based on how the intervention is perceived by pregnant women (assessed using a 5-point Likert scale : higher score mean a better outcome)

SECONDARY OUTCOMES:
Functional disability | Baseline (Pre-intervention) and week 16 (Post-intervention)
  Assessed using the Pelvic Girdle Questionnaire (PGQ) (score range from 0 (minimum) to 75 (maximum) : higher score mean a worst outcome)
Fear avoidance behaviors | Baseline (Pre-intervention) and week 16 (Post-intervention)
  Assessed using the Tampa Scale of Kinesiophobia (TSK) (score range from 17 (minimum) to 68 (maximum) : higher score mean a worst outcome)
Level of anxiety | Baseline (Pre-intervention) and week 16 (Post-intervention)
  Assessed using the State-Trait Anxiety Inventory (STAI) (score range from 20 (minimum) to 80 (maximum) : higher score mean a worst outcome)
Depression | Baseline (Pre-intervention) and week 16 (Post-intervention)
  Assessed using the Beck Depression Inventory (BDI) (score range from 0 (minimum) to 63 (maximum) : higher score mean a worst outcome)
Physical activity levels | Baseline (Pre-intervention) and week 16 (Post-intervention)
  Assessed using the Pregnancy Physical Activity Questionnaire (PPAQ) (weekly energy expenditure (MET-h·week-1), score range from 0 (minimum) to 1631 (maximum) : higher score mean a more active person)
Lumbopelvic pain (incidence and frequency) | Baseline (Pre-intervention)
  Defined as a weekly self-reported incidence and frequency of lumbopelvic pain (determined based on the number of episode)
Lumbopelvic pain (incidence and frequency) | 16 weeks follow-up
  Defined as a weekly self-reported incidence and frequency of lumbopelvic pain (determined based on the number of episode)
Lumbopelvic pain (incidence and frequency) | Week 16 (Post-intervention)
  Defined as a weekly self-reported incidence and frequency of lumbopelvic pain (determined based on the number of episode)
Lumbopelvic pain (intensity) | Baseline (Pre-intervention)
  Defined as a weekly self-reported intensity of lumbopelvic pain using a 100 millimeters visual analog scale
Lumbopelvic pain (intensity) | 16 weeks follow-up
  Defined as a weekly self-reported intensity of lumbopelvic pain using a 100 millimeters visual analog scale
Lumbopelvic pain (intensity) | Week 16 (Post-intervention)
  Defined as a weekly self-reported intensity of lumbopelvic pain using a 100 millimeters visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Martin Descarreaux, DC, PhD, Study Director — Université du Québec à Trois-Rivières
Locations (1):
- Université du Québec à Trois-Rivières, Trois-Rivières, Quebec, Canada

REFERENCES:
- [Derived] Daneau C, Marchand AA, Bussieres A, O'Shaughnessy J, Ruchat SM, Descarreaux M. Effects of a motor control exercise program on lumbopelvic pain recurrences and intensity in pregnant women with a history of lumbopelvic pain: a study protocol for a randomized controlled feasibility trial. Pilot Feasibility Stud. 2022 Mar 21;8(1):65. doi: 10.1186/s40814-022-01024-0. PMID 35313988